CLINICAL TRIAL: NCT05737225
Title: The Effect of Regional Anesthesia Method on Tissue Oxygenation in Patients Who Will Undergo Percutaneous Transluminal Angioplasty
Brief Title: Regional Anesthesia for Percutaneous Transluminal Angioplasty
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Demet Coşkun, Prof. Dr., Gazi University
Other Study IDs: 775 (24.10.2022)
Record Dates: First submitted 2023-02-03; First posted 2023-02-21 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Peripheral Artery Occlusive Disease; Percutaneous Transluminal Angioplasty
Keywords: percutaneous transluminal angioplasty; tissue oxygenation
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1 | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Popliteal sciatic nerve block group: regional anesthesia applied patients who will undergo percutaneous transluminal angioplasty (PTA) procedure
  Interventions: Device: Near Infrared Spectroscopy (NIRS)
- Control group: patients who will undergo percutaneous transluminal angioplasty (PTA) procedure
  Interventions: Device: Near Infrared Spectroscopy (NIRS)

INTERVENTIONS:
Device: Near Infrared Spectroscopy (NIRS) — We will place Near Infrared Spectroscopy (NIRS) electrode on the foot to evaluate regional tissue oxygen saturation in both lower extremities before the performing regional anesthesia (popliteal sciatic nerve block) and then during the procedure.

SUMMARY:
In this study, the effects of regional anesthesia method applied in patients who will undergo percutaneous transluminal angioplasty for lower extremity revascularization will be investigated comparatively.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 18 years
* Peripheral artery occlusive disease
* Eligibility for PTA

Exclusion Criteria:

* Patients' refusal
* Under the age of 18
* Language problems (not knowing turkish)
* Psychological or mental disorders.
* Disturbance of Conscious level.
* Uncooperative patients
* Those who are allergic to anesthetic drugs to be used
* Those with contraindications for the application of peripheral nerve block (coagulopathy, skin infection at the block site)
* need for endotracheal intubation or general anesthesia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ASA I-III patients over the age of 18 who have been decided to perform elective PTA as a treatment method for peripheral arterial disease will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-09-24 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Tissue Oxygenation | During procedure
  Tissue oxygenation will be measured from both lower extremities by Near Infrared Spectroscopy for 30 min after popliteal sciatic nerve block and during procedure.

SECONDARY OUTCOMES:
Body Temperature of Lower Extremities | During procedure
  Body temperature will be measured simultaneously at 0-5-10-15-20-25 and 30th minutes after the application of the popliteal sciatic nerve block
Patient Satisfaction Score | 15 minutes after procedure
  Self-administrated satisfaction score will be collected with scale from 0 to 5. A score of "0" means extremely dissatisfied and that a score of "5" means extremely satisfied.
Surgeon Satisfaction Score | 15 minutes after procedure
  Self-administrated satisfaction score will be collected with scale from 0 to 5. A score of "0" means extremely dissatisfied and that a score of "5" means extremely satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No